CLINICAL TRIAL: NCT05649605
Title: Early Mental Response to Hormonal Treatment in Transgender Men - The EMRE Study
Brief Title: Early Mental Response - The EMRE Study
Acronym: EMRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Mats Holmberg, Chief Physician, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2019-004349-34 SE
Record Dates: First submitted 2022-11-04; First posted 2022-12-14 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Gender Dysphoria; Gender Identity; Gender Issues
MeSH Terms: conditions — Gender Dysphoria; Sexism | interventions — testosterone undecanoate; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, placebo controlled, double blind study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participating research staff will be blinded to the treatment the patient is receiving. The drug and placebo will be labelled by Tamro AB, which will ensure that Nebido and placebo cannot be separated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active comparator arm (Active Comparator): Active treatment
  Interventions: Drug: Testosterone treatment
- Placebo comparator arm (Placebo Comparator): Placebo treatment
  Interventions: Other: Placebo treatment

INTERVENTIONS:
Drug: Testosterone treatment — Cross-sex hormone therapy consisting of intramuscular injection of testosterone undecanoate 250mg/ml. 4ml (total dosage of 1000mg) administered by trained nurse in the gluteal region at visit 1.
  Other Names: Nebido (3-oxandrostenderivate), testosterone undecanoate
  Arms: Active comparator arm
Other: Placebo treatment — Saline solution. Intramuscular injection of physiological saline solution. 4ml administered by trained nurse in the gluteal region at visit 1.
  Other Names: Sodium chloride solution
  Arms: Placebo comparator arm

SUMMARY:
Primary question: Does transgender men's experience of gender incongruence improve within 6 weeks of hormonal treatment compared to placebo? Long before any bodily changes occur.

Secondary question: Does transgender men´s experience of self-esteem, quality of life, sexual desire, aggression, depression/anxiety, impulsiveness, and emotional reactivity improve during 6 weeks of cross-sex hormone therapy compared to placebo? Gender dysphoria is a condition characterized by a perceived incongruence between the body and identity. For several decades this condition has been treated with cross-sex hormone therapy and surgery, among others, in order to change the body to be more congruent with the perceived gender identity. Patient satisfaction with this treatment is very high where an overwhelming majority of patients live the rest of their lives according to their perceived gender. A clinical observation, however, is that most patients experience that the congruence between the perceived gender and the assigned one improves very quickly on hormonal treatment. Long before any changes to the body have taken place. This may be partly due to relief from having finally started treatment (i.e. a psychological/social explanation) but an alternative (and much more likely) explanation is that the hormonal treatment directly affects the brain. Since the cause of gender dysphoria is unknown today, this study is therefore a step in trying to clarify the mechanism. In addition, it is of value to be able to demonstrate the benefits of hormonal treatment in these patients. Finally, there is a basic research motive for this study. The effect of sex hormones on the brain is very well known from a clinical perspective but all the more unknown from a research perspective. This study will contribute knowledge in this area.

DETAILED DESCRIPTION:
1.1 Gender dysphoria (GD) is currently a psychiatric diagnosis in Sweden. To meet the criteria according to the International Classification of Diseases (ICD-10), the patient must demonstrate a strong and persistent cross-gender identification coupled with persistent discomfort with his or her sex. ICD-10 uses the term "transsexualism" rather than "gender dysphoria". For the purpose of this study, we limit ourselves to adult transgender men by defining transsexualism in accordance with the diagnostic criteria for ICD-10.

GD is associated with significant suffering, reduced quality of life, and high self-reported disabilities. Comorbidity with other psychiatric diagnoses is high and the condition is linked to minority stress and discrimination.

1.2 Gender-confirming hormone therapy Cross-sex hormone therapy (CHT) is in most cases an important part of gender-confirming care of binary trans people. In trans men (assigned women at birth), CHT usually consists of testosterone alone. The method of administration is either topical gel or intramuscular injection. In this study, subjects are consequently treated with testosterone through intramuscular injection.

1.3 Effects of estradiol on the brain Estradiol is the predominant estrogen used as part of CHT in trans women. In trans men, the total levels of estradiol are lowered to levels equivalent to those of cis-men through negative feedback from testosterone administration. Estradiol is a steroid hormone that diffuses easily across the cell membrane and the blood-brain barrier (BBB), thus affecting the brain.

Sudden falls in estradiol concentrations and persistent estradiol deficiency are linked to mood swings. A suggested cause is estradiol's effect on dopaminergic, cholinergic, Gamma-aminobutyric acid (GABA) ergic, glutamatergic and serotonergic neurotransmission. Estradiol increases serotonin levels and other monoamines in the synapse by affecting monoamine oxidase and intraneuronal serotonin transport activity. It has also been suggested to increase binding sites in areas of the brain relevant to mood and cognition, and to increase binding to the serotonin 2A receptor - the most common serotonin receptor in the brain.

1.4 Effects of testosterone on the brain Testosterone is a steroid hormone that diffuses easily across the BBB and the cell membrane. Effects are mediated mainly via the androgen receptor (AR).

Testosterone can affect target cells directly or through conversion to the more potent form of dihydrotestosterone (DHT), or via conversion to estradiol. Both testosterone and DHT act directly on the AR, but DHT has a higher affinity for it. The enzymes that mediate the conversion of testosterone to DHT or estradiol (5-alpha-reductase and aromatase, respectively) vary between different tissues. Aromatase is abundant in parts of the Central Nervous System (CNS), suggesting that the effects of testosterone can be mediated through conversion to estradiol.

Serotonin plays a central role in mood, stress regulation, and cognition. Testosterone affects serotonin signaling, although serotonergic neurons do not express androgen receptors. A Positron Emission Tomography (PET) study showed that serum testosterone levels correlate with a proxy measure of serotonin tone in healthy men, suggesting that men with high serum testosterone have a higher serotonergic tone. However, the clinical relevance of this is unclear.

Several studies show that testosterone plays an important role in sexual desire, sexual thoughts, and sexual activity in men. The correlation between testosterone and aggression has been thoroughly studied. Physically and verbally aggressive behavior has been suggested to correlate with high levels of plasma testosterone while moderate supraphysiological levels show no change in aggression.

Several studies suggest a link between depression and hypogonadism in men. The conditions share symptoms such as depression, fatigue, decreased libido, decreased energy, and decreased general joy in life. Lower testosterone levels have been found in depressed men compared to healthy controls and these symptoms can be mitigated with testosterone treatment. In addition to depression, the correlations between several other mental illnesses and abnormal levels of testosterone have been studied. Low levels have been found in schizophrenia and chronic sleep disorders. High levels have been found in post-traumatic stress and have been associated with low stress tolerance in young men. Improvement of obsessive-compulsive disorder with antiandrogen therapy has been reported, as well as increased severity of Tourette-related symptoms with testosterone therapy.

1.5 Mental effects of hormonal therapy in trans men Specifically in trans men, increased sexual desire after CHT has been reported. Whether these changes are due to hormone therapy or the fact that starting treatment is seen as a period of joy after an often long investigation period is not known. Decreased sensitivity/sensitivity after hormone insertion has also been reported. A clinical observation is that patients experience a marked improvement in their gender incongruence already after a short period of CHT (i.e. long before any changes in the body occurred).

2. Risk-benefit evaluation The cause of GD is today basically unknown. The condition is mainly considered congenital where abnormal development of the brain during the time gender identity and phenotype develops is a theory. Clinically, this condition has been treated for several decades with an adaptation of the body to the perceived identity with the help of CHT and surgery. Patient satisfaction with this treatment is high and an overwhelming majority live the rest of their lives as the perceived gender.

This study is important from a variety of perspectives. Partly regarding the question of what causes the actual condition of gender incongruence, partly regarding the efficacy of the actual treatment, and finally partly from a basic research perspective where many of the sex hormones' effects on the brain are poorly researched.

The benefit is thus great with this study. Performing randomized, placebo-controlled studies on the trans group have long been considered impossible. However, thanks to the fact that this study has been planned in consultation with transgender people, a design has been constructed that enables comparison with placebo.

In terms of risks, patients receive an injection of Nebido (4ml/1000mg) or placebo. This is standard clinical treatment and when it is time for syringe number two (after six weeks), the study ends and the placebo group will then receive Nebido accordingly to clinical routine.

Risks with the injection are well known. The injection can cause local pain and a slight cough, they are both transient.

3. Objectives: The aim of this study is to capture and describe the early effects on the brain of CHT in trans men.

3.1 Primary aim: The primary purpose of this study is to study whether treatment with testosterone provides greater improvement in the experience of gender incongruence compared to placebo in trans men.

3.2 Secondary aim: The secondary purpose of this study is to examine changes in self-esteem, quality of life, sexual desire, aggression, depression/anxiety, impulsiveness, and emotional reactivity during the first six weeks of hormonal treatment compared to placebo.

3.3 Primary variable: The difference in points on the Transgender Congruence Scale between inclusion, after two weeks of treatment and after six weeks of treatment with testosterone or placebo.

3.4 Secondary variable: The difference in points on Rosenberg Self-Esteem Scale, Brunnsviken Brief Quality of Life Scale, Sexual Desire Inventory, Buss-Perry Aggression Questionnaire, Montgomery Asberg Depression Rating Scale, Barratt Impulsiveness Scale, and Perth Emotional Reactivity Scale-Short form between inclusion, after two weeks of treatment and after 6 weeks of treatment with testosterone or placebo.

4. Study design and Procedures

4.1 Overall study design This is a prospective, randomized, double-blind placebo-controlled study of 70 individuals with assigned female sex at birth and recently diagnosed with transsexualism according to ICD-10 (F64.0). The diagnosis of transsexualism is made by a psychiatrist, after which the patient is referred to an endocrinologist who makes his own assessment of the suitability for CHT.

There is a long, well-established clinical treatment for these patients with testosterone.

In the study, participants are treated with testosterone (Nebido) in standard dosage according to Summary of Product Characteristics (SmPC) or placebo, both in injection form. Nebido treatment is started with two injections six weeks apart and every 12 weeks thereafter. To minimize deviations from clinical routine, the study length has therefore been set at six weeks, after which all patients are offered continued treatment according to clinical routine.

4.2 Procedures and flow chart Se procedures and flow chart pdf provided in the "Document section".

4.3 Biological sampling procedures

4.3.1 Handling, storage, and destruction of biological samples Sampling for safety and efficacy monitoring is performed according to standard at ANOVA before inclusion (before drug administration). The following assays include S-Testosterone, S-Estradiol, S-Luteinising Hormone (LH), S-Follicle Stimulating Hormone (FSH), S-Sex Hormone Binding Globulin (SHBG), P-Aspartate aminotransferase (ASAT), P-Alanine Aminotransferase (ALAT), S-25-OH-Vitamin D, B-Hemoglobin (Hb), B-Erythrocyte Volume Fraction (EVF), B-Mean Concentration Hemoglobin (MCH), B-Mean Corpuscular Hemoglobin Concentration (MCHC), B-Leukocyte Particle Concentration (LPK), B-Thrombocyte Particle Concentration (TPK), P-Calcium, P-C-Reactive protein (CRP), P-Phosphate, fasting S-Insulin, P-Glucose, P-Gamma-glutamyl Transferase (GGT), B-HemoglobinA1c, P-High-density lipoprotein (HDL), fasting P-Low-density lipoprotein (LDL), fasting P-Cholesterol, fasting P-Triglyceride, P-Sodium, S-Prolactine, S-free Triiodothyronine (T3), S-free Thyroxine (T4) and S-Thyroid-Stimulating Hormone (TSH). After 6 weeks of treatment, S-Testosterone, S-Estradiol, S-LH, S-FSH, S-SHBG are checked. All samples are analyzed at Karolinska University Hospital Laboratory. No samples are saved.

4.3.2 Total volume blood per study subject The total volume of blood taken from each study subject during the study is a maximum of 40 ml.

4.4 Study end The study ends when the last researcher has completed the last follow-up (LSLV).

The study may be terminated prematurely if it turns out that the treatment causes a large number of unwanted serious events or if the recruitment of research personnel cannot be fulfilled within a reasonable time limit. If the study is terminated prematurely, or temporarily stopped, the investigator shall immediately inform the researchers of this and ensure appropriate treatment and follow-up. The regulatory authority should be informed as soon as possible, but no later than within 15 days.

Decision on early termination of the study is made by the sponsor.

ELIGIBILITY:
Inclusion criteria:

1. Well-informed written consent to participate in the study.
2. Transgender man given the ICD-10 diagnosis of transsexualism.
3. A desire for complete gender-confirming hormonal treatment.
4. Approved for Nebido treatment by a clinically responsible Endocrinologist.

Exclusion criteria:

1. A concomitant hormonal condition affecting the gonadal axis (e.g. Congenital Adrenal Hyperplasia, Poly Cystic Ovary Syndrome, Complete Androgen Insensitivity Syndrome, Partial Androgen Insensitivity Syndrome, untreated thyroid disease, untreated hypercortisolism, etc.).
2. A disability that prevents the patient from fully participating in the study.
3. Treatment with steroid hormones (androgens, estrogens, progestogens, or continuous treatment with oral corticosteroids within the last three months).
4. Previous use of hormone preparations without a doctor's prescription.
5. Laboratory samples significantly outside the normal reference range.
6. Anamnestic or investigational suspicion of breast cancer or existing or previous liver tumors.
7. Levels of P-ASAT, P-ALAT, or P-GT at the screening time that are> 2 times the reference range.
8. Hypersensitivity to the active substance or to any of the excipients.
9. Ongoing pregnancy or wishes for a pregnancy in the near future.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender males
Enrollment: 70 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in baseline gender incongruence at 2 and 6 weeks respectively | Performed at visit 2 (pre treatment), 2 weeks into treatment (performed at distance) and after 6 weeks of treatment (visit 3, study ends).
  Score according to Transgender Congruence Scale. The total score ranges from a mean value of 12 items scored from 1 to 5. The mean value ranges from 1 to 5 points in total. A low score indicates a high level of gender dysphoria and a high score indicates a low level of gender dysphoria.

SECONDARY OUTCOMES:
Changes in baseline slef-esteem at 2 and 6 weeks respectively. | Performed at visit 2 (pre treatment), 2 weeks into treatment (performed at distance) and after 6 weeks of treatment (visit 3, study ends).
  Scores according to Rosenberg self-esteem scale. The scale contains 10 items scored from 0 to 3 points. Total score ranges from 0-30 points. High scores indicate a high self-esteem and low scores indicate a low self-esteem.
Changes in baseline quality of life at 2 and 6 weeks respectively. | Performed at visit 2 (pre treatment), 2 weeks into treatment (performed at distance) and after 6 weeks of treatment (visit 3, study ends).
  Scores according to Brunnsviken Brief Quality of Life Inventory. The scale contains 12 items scored from 0 to 4. The total score ranges from 0 to 96 points. A low score indicates a low quality of life and a high score indicates a high quality of life.
Changes in baseline sexual desire at 2 and 6 weeks respectively. | Performed at visit 2 (pre treatment), 2 weeks into treatment (performed at distance) and after 6 weeks of treatment (visit 3, study ends).
  Scores according to Sexual Desire Inventory. The scale contains 13 items in total. Items are scored from 0 to 5. Total score ranges from 0 to 101 points measuring total sexual desire. Items 1 to 9 contains a subscale measuring dyadic sexual desire. Items 10 to 13 contains a subscale measuring solitary sexual desire. A low score indicates a low sexual desire and a high score indicates a high sexual desire on both the main scale and subscales.
Changes in baseline aggression at 2 and 6 weeks respectively. | Performed at visit 2 (pre treatment), 2 weeks into treatment (performed at distance) and after 6 weeks of treatment (visit 3, study ends).
  Scores according to Buss-Perry Aggression Questionnaire. The scale contains 29 items in total scored from 1 to 5. Total score ranges from 29 to 145. The scale includes 4 subscales. Physical Aggression (items 1-9), verbal Aggression (items 10-14), anger (items 15-21), and hostility (items 22-29). A high score indicates high aggression and a low score indicates low aggression on both the main scale and subscales.
Changes in baseline depressive symptoms and anxiety at 2 and 6 weeks respectively. | Performed at visit 2 (pre treatment), 2 weeks into treatment (performed at distance) and after 6 weeks of treatment (visit 3, study ends).
  Scores according to Montgomery Asberg Depression Rating Scale.The scale contains 9 items scored from 0 to 6. Total score ranges from 0 to 54. 0 to12 indicates no or mild depression. 13 to 19 points indicate mild depression. 20 to 34 indicate mild depression. 35 to 54 indicate severe depression.
Changes in baseline impulsiveness at 2 and 6 weeks respectively. | Performed at visit 2 (pre treatment), 2 weeks into treatment (performed at distance) and after 6 weeks of treatment (visit 3, study ends).
  Scores according to Barratt Impulsiveness Scale. The scale contains 30 items scored from 1 to 4. Total score ranges from 30 to 120. The scale contains 3 subscales. Attentional scale with a total of 8 items (divided in two - attention and cognitive instability, 5 and 3 items respectively). Motor scale with a total of 11 items (divided in two - attention and cognitive instability, 7 and 4 items respectively). Non-planning scale (divided in two - self-control and cognitive complexity, 6 and 5 items respectively). A high score indicates a high impulsiveness and a low score indicates a low impulsiveness on all scales.
Changes in baseline emotional reactivity at 2 and 6 weeks respectively. | Performed at visit 2 (pre treatment), 2 weeks into treatment (performed at distance) and after 6 weeks of treatment (visit 3, study ends).
  Scores according to Perth Emotional Reactivity Scale-Short Form. The scale contains 18 items scored from 1 to 5. Total score ranges from 18 to 90. The scale contains 8 sub scales. Negative-activation-scale, sum total score from items 2, 8, 14. Negative-intensity-scale, sum total score from items 6, 12, 18. Negative-duration-scale, sum items 4, 10, 16. Positive-activation-scale, sum total score from items 1, 7, 13. Positive-intensity-scale, sum total score from items 5, 11, 17. Positive-duration-scale, sum total score from items 3, 9, 15. General negative reactivity-scale, sum total score from all even numbered items. General positive reactivity-scale, sum total score from all odd numbered items. A high score indicates a high emotional reactivity and a low score indicates a low emotional reactivity on all scales.

CONTACTS AND LOCATIONS:
Overall Officials: Mats Holmberg, MD. PhD., Principal Investigator — ANOVA Karolinska sjukhuset
Locations (1):
- Karolinska Universitetssjukhuset, ANOVA, Stockholm, Sweden

REFERENCES:
- [Background] Mahfouda S, Moore JK, Siafarikas A, Hewitt T, Ganti U, Lin A, Zepf FD. Gender-affirming hormones and surgery in transgender children and adolescents. Lancet Diabetes Endocrinol. 2019 Jun;7(6):484-498. doi: 10.1016/S2213-8587(18)30305-X. Epub 2018 Dec 6. PMID 30528161
- [Background] de Vries AL, McGuire JK, Steensma TD, Wagenaar EC, Doreleijers TA, Cohen-Kettenis PT. Young adult psychological outcome after puberty suppression and gender reassignment. Pediatrics. 2014 Oct;134(4):696-704. doi: 10.1542/peds.2013-2958. Epub 2014 Sep 8. PMID 25201798
- [Background] Frisen L, Soder O, Rydelius PA. [Dramatic increase of gender dysphoria in youth]. Lakartidningen. 2017 Feb 22;114:EFMY. Swedish. PMID 28245038
- [Background] American Psychiatric association. Diagnostic and statistical manual of mental disorders, 5th edition (DSM-5). Arlington VA; 2013.
- [Background] World Health Organization. International statistical classification of diseases and related health problems, 10th revision (ICD-10). Geneva; 1992.
- [Background] World Professional Association for Transgender Health (WPATH). Standards of Care for the Health of Transsexual, Transgender, and Gender Nonconforming People (7th version). 2009.
- [Background] Socialstyrelsen. God vård av vuxna med könsdysfori. 2015.
- [Background] Hembree WC, Cohen-Kettenis P, Delemarre-van de Waal HA, Gooren LJ, Meyer WJ 3rd, Spack NP, Tangpricha V, Montori VM; Endocrine Society. Endocrine treatment of transsexual persons: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2009 Sep;94(9):3132-54. doi: 10.1210/jc.2009-0345. Epub 2009 Jun 9. PMID 19509099
- [Background] Gijs L, Brewaeys A. Surgical Treatment of Gender Dysphoria in Adults and Adolescents: Recent Developments, Effectiveness, and Challenges. Annu Rev Sex Res. Taylor & Francis; 2007 Mar 1;18(1):178-224.
- [Background] Smith YL, Van Goozen SH, Kuiper AJ, Cohen-Kettenis PT. Sex reassignment: outcomes and predictors of treatment for adolescent and adult transsexuals. Psychol Med. 2005 Jan;35(1):89-99. doi: 10.1017/s0033291704002776. PMID 15842032
- [Background] Davy Z. The DSM-5 and the Politics of Diagnosing Transpeople. Arch Sex Behav. 2015 Jul;44(5):1165-76. doi: 10.1007/s10508-015-0573-6. PMID 26054486
- [Background] Zeluf G, Dhejne C, Orre C, Nilunger Mannheimer L, Deogan C, Hoijer J, Ekeus Thorson A. Health, disability and quality of life among trans people in Sweden-a web-based survey. BMC Public Health. 2016 Aug 30;16(1):903. doi: 10.1186/s12889-016-3560-5. PMID 27576455
- [Background] Collin L, Reisner SL, Tangpricha V, Goodman M. Prevalence of Transgender Depends on the "Case" Definition: A Systematic Review. J Sex Med. 2016 Apr;13(4):613-26. doi: 10.1016/j.jsxm.2016.02.001. Epub 2016 Mar 25. PMID 27045261
- [Background] Bockting W, Knudson G, Goldberg JM, Goldberg J, Lindenberg D, Hunt R, et al. Counselling and Mental Health Care of Transgender Adults and Loved Ones. 2006.
- [Background] Newfield E, Hart S, Dibble S, Kohler L. Female-to-male transgender quality of life. Qual Life Res. 2006 Nov;15(9):1447-57. doi: 10.1007/s11136-006-0002-3. Epub 2006 Jun 7. PMID 16758113
- [Background] Pfäfflin F, Junge A. Thirty years of international follow-up studies after sex reassignment surgery: a comprehensive review 1961-1991. 1998.
- [Background] Läkemedelsindustriföreningen. Androcur [Internet]. Fass. 2018. Available from: https://www.fass.se/LIF/product?userType=0&nplId=19780414000015
- [Background] McEwen BS, Alves SE. Estrogen actions in the central nervous system. Endocr Rev. 1999 Jun;20(3):279-307. doi: 10.1210/edrv.20.3.0365. No abstract available. PMID 10368772
- [Background] Kuhl H. Pharmacology of estrogens and progestogens: influence of different routes of administration. Climacteric. 2005 Aug;8 Suppl 1:3-63. doi: 10.1080/13697130500148875. PMID 16112947
- [Background] Douma SL, Husband C, O'Donnell ME, Barwin BN, Woodend AK. Estrogen-related mood disorders: reproductive life cycle factors. ANS Adv Nurs Sci. 2005 Oct-Dec;28(4):364-75. doi: 10.1097/00012272-200510000-00008. PMID 16292022
- [Background] Champe PC, Harvey RA, Ferrier DR. Biochemistry. 4th ed. Baltimore; 2008.
- [Background] Wang C, Liu Y, Cao JM. G protein-coupled receptors: extranuclear mediators for the non-genomic actions of steroids. Int J Mol Sci. 2014 Sep 1;15(9):15412-25. doi: 10.3390/ijms150915412. PMID 25257522
- [Background] Banks WA. Brain meets body: the blood-brain barrier as an endocrine interface. Endocrinology. 2012 Sep;153(9):4111-9. doi: 10.1210/en.2012-1435. Epub 2012 Jul 9. PMID 22778219
- [Background] Cyr M, Calon F, Morissette M, Grandbois M, Di Paolo T, Callier S. Drugs with estrogen-like potency and brain activity: potential therapeutic application for the CNS. Curr Pharm Des. 2000 Aug;6(12):1287-312. doi: 10.2174/1381612003399725. PMID 10903393
- [Background] Perfalk E, Cunha-Bang SD, Holst KK, Keller S, Svarer C, Knudsen GM, Frokjaer VG. Testosterone levels in healthy men correlate negatively with serotonin 4 receptor binding. Psychoneuroendocrinology. 2017 Jul;81:22-28. doi: 10.1016/j.psyneuen.2017.03.018. Epub 2017 Mar 22. PMID 28426945
- [Background] Nieschlag E, Behre HM. Testosterone: action, deficiency, substitution. 4th ed. Cambridge: Cambridge University Press; 2012.
- [Background] Zarrouf FA, Artz S, Griffith J, Sirbu C, Kommor M. Testosterone and depression: systematic review and meta-analysis. J Psychiatr Pract. 2009 Jul;15(4):289-305. doi: 10.1097/01.pra.0000358315.88931.fc. PMID 19625884
- [Background] Rohr UD. The impact of testosterone imbalance on depression and women's health. Maturitas. 2002 Apr 15;41 Suppl 1:S25-46. doi: 10.1016/s0378-5122(02)00013-0. PMID 11955793
- [Background] Defreyne J, Elaut E, Kreukels B, Fisher AD, Castellini G, Staphorsius A, Den Heijer M, Heylens G, T'Sjoen G. Sexual Desire Changes in Transgender Individuals Upon Initiation of Hormone Treatment: Results From the Longitudinal European Network for the Investigation of Gender Incongruence. J Sex Med. 2020 Apr;17(4):812-825. doi: 10.1016/j.jsxm.2019.12.020. Epub 2020 Jan 31. PMID 32008926
- [Background] Pope HG Jr, Cohane GH, Kanayama G, Siegel AJ, Hudson JI. Testosterone gel supplementation for men with refractory depression: a randomized, placebo-controlled trial. Am J Psychiatry. 2003 Jan;160(1):105-11. doi: 10.1176/appi.ajp.160.1.105. PMID 12505808

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT05649605/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-20): https://cdn.clinicaltrials.gov/large-docs/05/NCT05649605/ICF_001.pdf